CLINICAL TRIAL: NCT05545475
Title: Safety of Anticoagulant Therapy After Tissue Glue for Gastric Varices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Taian City Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20220117-Qilu
Record Dates: First submitted 2022-02-23; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-01

CONDITIONS: Anticoagulants and Bleeding Disorders; Tissue Adhesion; Gastric Varices Bleeding
Keywords: anticoagulants; tissue glue; gastric varices
MeSH Terms: conditions — Hemostatic Disorders; Tissue Adhesions; Esophageal and Gastric Varices | interventions — Heparin, Low-Molecular-Weight; Nadroparin; Warfarin; Enoxaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anticoagulation group: 1 mg/kg of nadroparin calcium or enoxaparin every 12 h, 5000 IU of low molecular weight heparin (LMWH) every 12 h, 20 mg of rivaroxaban once daily, or warfarin adjusted by an increase or decrease of 0.75 mg until the target international normalized ratio (INR) of 2-3 was reached.
  Interventions: Drug: Low molecular weight heparin
- Control group: No anticoagulation group.

INTERVENTIONS:
Drug: Low molecular weight heparin — Anticoagulants were given. When using warfarin, international normalized ratio (INR) was detected every 3-4 days and adjusted carefully by 0.75mg dosage until achieve the target level of 2-3.
  Other Names: Nadroparin calcium; Rivaroxiban; Warfarin; Enoxaparin
  Groups: Anticoagulation group

SUMMARY:
This study aimed to clarify the safety of anticoagulant therapy after glue injection for cirrhotic variceal bleeding patients with portal vein thrombosis.

DETAILED DESCRIPTION:
Acute esophagogastric varices bleeding is a common gastroenterological emergency. And the bleeding from ruptured gastric varices is massive and difficulty to stop, even after aggressive pharmacological and conservative treatment. Even after aggressive pharmacological and conservative treatment, maintaining patients without bleeding for a long time is still a challenging clinical problem. Endoscopic tissue adhesive injection is recommended by many international guidelines for acute hemostasis and secondary prevention of gastric variceal bleeding. However, postoperative glue extrusion is inevitable, and the the rebleeding caused by glue ulcers is a problem that is often faced in clinical work. In patients with portal vein thrombosis, the need for anticoagulation and the choice of anticoagulant drugs need to be carefully evaluated in terms of risk and benefit, as the dual conflicts of thrombosis and anticoagulation are involved. At present, there is no in-depth study or consensus on the effect of anticoagulation on rebleeding after glue injection in patients with portal vein thrombosis. This study is of great significance for the treatment and prognosis of patients with gastric varices combined with portal vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cirrhosis
* Portal hypertension with gastric varices
* diagnosis of PVT by imaging examination
* undergo glue injection for gastric varices

Exclusion Criteria:

* hepatocellular carcinoma or other extrahepatic malignancy
* isolated portal cavernoma
* treatment with TIPS, thrombolysis, thrombectomy or liver transplantation
* previous long-term anticoagulation therapy for various reasons
* pregnant women
* previous endoscopic treatment of GVs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cirrhotic patients complicated with imaging-confirmed PVT and undergoing injection of tissue adhesive for GVs from three tertiary referral hospitals (Qilu Hospital of Shandong University, Shandong Provincial Hospital, and Taian City Central Hospital) were screened.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-18 (Estimated); Study Completion 2024-01-18 (Estimated)

PRIMARY OUTCOMES:
the incidence of a bleeding episode from glue cast extrusion | 6-month
  hematemesis, melena, or a ≥ 2 g drop in hemoglobin, with endoscopy-confirmed active spurting or oozing from the site of extrusion of glue casts, or an ulcer with an adherent clot or a visible vessel and no other sources of bleeding

SECONDARY OUTCOMES:
death | 6-month
  death from all causes of illness related to liver dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao, PhD., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China